CLINICAL TRIAL: NCT02640313
Title: Molecular Imaging of Plaque Vulnerability Using 18F-choline PET-MRI in Carotid Artery Atherosclerosis Patients
Brief Title: Molecular Imaging of Plaque Vulnerability
Acronym: PARISK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL43466.068.13/ABR43466; NCT01899014 (obsolete NCT alias)
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Plaque, Atherosclerotic
Keywords: 18F-fluormethylcholine; [F18] choline; [F18] fluormethylcholine
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-choline PET-MR imaging (Experimental): Intervention: 18F-choline PET-MR imaging.
  Drug: 18F-choline, dosis 4 MBq/kg body-weight (maximum 360 MBq), administered intravenously as a single dose.
  Procedure: dynamic and static 18F-choline PET-MR.
  Interventions: Drug: 18F-choline PET-MR imaging

INTERVENTIONS:
Drug: 18F-choline PET-MR imaging — Dynamic and static 18F-choline PET-MR imaging
  Other Names: PET-MRI

SUMMARY:
Accumulating data in the literature suggests that radiolabeled-choline (18F-choline) is a sensitive molecular tracer for PET imaging that is taken up in activated cells and, as such, is able to identify active inflammatory sites. The investigators hypothesize that 18F-choline is also highly taken up in vulnerable plaques in comparison to the stable ones.

DETAILED DESCRIPTION:
Accumulation and subsequent activation of inflammatory cells in the atherosclerotic plaques play an essential role in transforming a stable plaque into a vulnerable plaque at risk to rupture. On this basis, the study aims to evaluate the diagnostic performance of 18F-choline PET in identifying ongoing inflammation within atherosclerotic plaques. The investigators hypothesize that 18F-choline PET is efficient in detecting intraplaque inflammation and identify vulnerable plaques that are prone to rupture in comparison to the stable ones.

It is likely that by correlating the inflammatory status of an atherosclerotic plaque (on 18F-choline PET) with the presence of other vulnerable plaque features (on MR imaging) would be of high clinical relevance for clinical diagnosis of vulnerable plaques.

ELIGIBILITY:
Inclusion Criteria:

* Patients known with symptomatic carotid artery stenosis (≥2 mm carotid plaque on duplex ultrasound), who are scheduled in the clinical setting to undergo a carotid endarterectomy or who are referred to conservative therapy;
* Age 18 years and older (no maximum age);
* Informed consent by signing informed consent form regarding this study.

Exclusion Criteria:

* Dementia, pregnancy, nursing mothers;
* Serious neurological deficits at symptomatic side (hemi paralysis, complete aphasia);
* Severe heart failure NYHA III-IV and severe pulmonary dysfunction dependent on oxygen supply;
* Patients with contra-indications for MRI (ferromagnetic implants like pacemakers or other electronic implants, metallic splinters in the eyes, vascular clips, claustrophobia, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
18F-choline uptake, as marker of plaque inflammation | 1 year
  • To assess on PET the uptake of 18F-choline tracer in the symptomatic carotid artery plaque, given as Target-to-Background uptake Ratio (TBR);
correlate the intra-plaque uptake of 18F-choline on PET with the total area of CD68-positivity within the symptomatic plaque | 1 year
  • In case of carotid surgery, to correlate the intra-plaque uptake of 18F-choline on PET with the total area of CD68-positivity within the symptomatic plaque, as a measure of plaque inflammation and vulnerability on histology
sensitivity, specificity, negative predictive value of 18F-choline PET | 1 year
  • To determine the sensitivity, specificity, negative predictive value of 18F-choline PET in diagnosis of vulnerable plaques.

SECONDARY OUTCOMES:
Correlation of F18-Choline uptake vs other histologic plaque parameters. | 1 year
  • In case of carotid surgery, to correlate the intra-plaque 18F-choline uptake on PET with other histologic plaque parameters besides inflammation, such as the total area of intra-plaque lipid core, haemorrhage, fibrous tissue and calcifications;
Correlation of F18-Choline uptake vs PET and MRI parameters of atherosclerotic plaque | 1 year
  • To correlate the intra-plaque 18F-choline uptake on PET and MRI parameters of atherosclerotic plaque, such as % of intra-plaque fibrous tissue, lipid core, hemorrhage, calcifications;
Correlation of F18-choline plaque uptake vs 18F-FDG uptake | 1 year
  • To correlate the intra-plaque 18F-choline uptake on PET with the already established FDG PET imaging parameters of atherosclerotic plaque, such as inflammation;
Symptomatic vs asymptomatic F18-Choline uptake | 1 year
  • To compare on PET the 18F-choline uptake in the symptomatic carotid plaque with the uptake in the asymptomatic contralateral carotid artery.
Correlation of F18choline plaque uptake vs cardiovascular risk profile | 1 year
  • To evaluate a possible association between the degree of 18F-choline uptake on PET with patients' cardiovascular risk profile and medical history.

CONTACTS AND LOCATIONS:
Overall Officials: M. Eline Kooi, PhD, Study Director — Maastricht University Medical Center; Jochem van der Pol, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bucerius J, Schmaljohann J, Bohm I, Palmedo H, Guhlke S, Tiemann K, Schild HH, Biersack HJ, Manka C. Feasibility of 18F-fluoromethylcholine PET/CT for imaging of vessel wall alterations in humans--first results. Eur J Nucl Med Mol Imaging. 2008 Apr;35(4):815-20. doi: 10.1007/s00259-007-0685-x. Epub 2008 Jan 6. PMID 18183393
- [Background] Forster S, Rominger A, Saam T, Wolpers S, Nikolaou K, Cumming P, Reiser MF, Bartenstein P, Hacker M. 18F-fluoroethylcholine uptake in arterial vessel walls and cardiovascular risk factors: correlation in a PET-CT study. Nuklearmedizin. 2010;49(4):148-53. doi: 10.3413/nukmed-0299. Epub 2010 Jun 8. PMID 20532464
- [Background] Kato K, Schober O, Ikeda M, Schafers M, Ishigaki T, Kies P, Naganawa S, Stegger L. Evaluation and comparison of 11C-choline uptake and calcification in aortic and common carotid arterial walls with combined PET/CT. Eur J Nucl Med Mol Imaging. 2009 Oct;36(10):1622-8. doi: 10.1007/s00259-009-1152-7. Epub 2009 May 9. PMID 19430785
- [Derived] Voo S, Kwee RM, Sluimer JC, Schreuder FH, Wierts R, Bauwens M, Heeneman S, Cleutjens JP, van Oostenbrugge RJ, Daemen JW, Daemen MJ, Mottaghy FM, Kooi ME. Imaging Intraplaque Inflammation in Carotid Atherosclerosis With 18F-Fluorocholine Positron Emission Tomography-Computed Tomography: Prospective Study on Vulnerable Atheroma With Immunohistochemical Validation. Circ Cardiovasc Imaging. 2016 May;9(5):e004467. doi: 10.1161/CIRCIMAGING.115.004467. PMID 27162131